CLINICAL TRIAL: NCT01491048
Title: Evaluation of Functional Rehabilitation Therapy in Patients Undergoing Physiotherapy After Total Hip Arthroplasty
Brief Title: Evaluation of Functional Rehabilitation in Patients Undergoing Physiotherapy After Total Hip Arthroplasty
Acronym: Artrhosis
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Hospital de Clinicas de Porto Alegre (Other)
Responsible Party: Principal Investigator, Carolina Sant'Anna Umpierres, Doctor Carolina Sant´Anna Umpierres, Hospital de Clinicas de Porto Alegre
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: 09242
Record Dates: First submitted 2011-10-30; First posted 2011-12-13 (Estimated); Last update posted 2011-12-13 (Estimated); Status verified 2011-12

CONDITIONS: Osteoarthritis, Hip
Keywords: Hip osteoarthritis; Physiotherapy; THA
MeSH Terms: conditions — Osteoarthritis, Hip | interventions — ORALIT; Papaverine; Physical Therapy Modalities; Tacrine

STUDY DESIGN:
Who Masked: Participant, Investigator
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- THA Physiotherapy (Active Comparator): Physiotherapy care during the period of hospitalization after THA.
  Interventions: Procedure: THA Physiotherapy; Procedure: No physiotherapy after THA
- No physiotherapy after THA (Active Comparator): No Physiotherapy care during the period of hospitalization after THA.
  Interventions: Procedure: No physiotherapy after THA

INTERVENTIONS:
Procedure: THA Physiotherapy — Patients will be randomized into two groups. The control group will receive care from the team of the THA Assistance Protocol already used by the HSG of HCPA without the intervention of physiotherapy. During hospitalization, the group of cases will be submitted to physical therapy associated with the intervention of the team of the THA Assistance Protocol.
  Other Names: osteoarthrosis, hip, physiotherapy.
  Arms: THA Physiotherapy
Procedure: No physiotherapy after THA — No physiotherapy after THA
  Other Names: Physiotherapy; THA

SUMMARY:
This study aims to objectively evaluate the implications of physiotherapeutic rehabilitation in the Assistance Protocol of Total Hip Arthroplasty (THA), by assessing the motor performance and testing the quality of life of patients undergoing THA surgery, to improve rehabilitation strategies for this population.

DETAILED DESCRIPTION:
The Total Hip Arthroplasty (THA) is a surgical procedure which has been used for more than half a century in the treatment of hip joint diseases.

The Physiotherapy is an important component in the care of patients undergoing THA.

In order to reduce the length of hospitalization after THA, to promote functional independence and to monitor clinical events during hospitalization and up to the 30th postoperative day, the Hip Surgery Group (HSG) of the Department of Orthopedics and Traumatology Department of Orthopedics and Traumatology of Hospital de Clinicas de Porto Alegre (HCPA) has developed a global, multidisciplinary Assistance Protocol of the HSG with outpatient consultations and scheduled home visits for patients that have undergone THA at HCPA.

The team which developed the Assistance Protocol of the HSG consists of orthopedic doctors and anesthesiologists, nurses and social workers.

The insertion of the Physiotherapist in the THA Assistance Protocol is of great importance owing to the professional skills of that professional in the areas of prevention and rehabilitation, working with the multidisciplinary team in functional evaluation and in physical therapy of patients that underwent THA.

The monitoring of the physiotherapist is essential to establish a functional diagnosis, aiming pain relief, promoting the early functional rehabilitation, the reintegration of the patients in their daily activities and offering a better quality of life through reintegration into social life.

ELIGIBILITY:
Inclusion Criteria:

* Patients with indication for THA.

Exclusion Criteria:

* Patients who refuse to participate in this study.
* Patients who live outside the city of Porto Alegre, due to difficulties for visits and the protocol monitoring.
* Patients with femoral neck fracture, due to the impossibility of evaluation.

Min Age: 18 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 104 (Actual)
Dates: Start 2009-07; Primary Completion 2011-10 (Actual); Study Completion 2011-10 (Actual)

PRIMARY OUTCOMES:
Physiotherapeutic Rehabilitation after THA. | 15 days after discharge
  Patients hospitalized in the HCPA for THA surgery, are submitted to an assessment and are randomized. Soon after, the treatment group receives the physiotherapy protocol while the control group receives guidance together with the THA Assistance Protocol. Fifteen days later the patients return to hospital where they are reassessed.

SECONDARY OUTCOMES:
Physiotherapeutic Rehabilitation after THA. | 15 days after discharge.
  Patients will be evaluated through tests of strength, range of motion, limb discrepancy, hip functionality and quality of life before and after discharge.

CONTACTS AND LOCATIONS:
Overall Officials: Carolina S Umpierres, Bachelor, Principal Investigator — Hospital de Clinicas de Porto Alegre
Locations (1):
- Hospital de Clinicas de Porto Alegre, Porto Alegre, Rio Grande do Sul, Brazil

REFERENCES:
- [Background] Walker RL, Fromm PO. Metabolism of iron by normal and iron deficient rainbow trout. Comp Biochem Physiol A Comp Physiol. 1976;55(4A):311-8. doi: 10.1016/0300-9629(76)90052-9. No abstract available. PMID 9242
- [Derived] Umpierres CS, Ribeiro TA, Marchisio AE, Galvao L, Borges IN, Macedo CA, Galia CR. Rehabilitation following total hip arthroplasty evaluation over short follow-up time: randomized clinical trial. J Rehabil Res Dev. 2014;51(10):1567-78. doi: 10.1682/JRRD.2014.05.0132. PMID 25856757